CLINICAL TRIAL: NCT06554626
Title: The Regimen of Blinatumomab and Venetoclax Sequenced With Inotuzumab Ozogamicin in Treating Precursor B Cell Acute Lymphoblastic Leukemia: A Phase II, Single Arm and Multicenter Study
Brief Title: Blinatumomab Plus Venetoclax Sequenced With Inotuzumab Ozogamicin in Treating B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240070C
Record Dates: First submitted 2024-08-06; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Precursor B-Cell Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dexamethasone; blinatumomab; venetoclax; Inotuzumab Ozogamicin; Methotrexate; pegaspargase; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Induction Cycle 1 and 2: Venetoclax for 2 weeks,oral; Blinatumomab for 2weeks, iv; Dexamethasone.
  Consolidation Cycle 3 and 5: Inotuzumab ozogamicin, iv. Cycle 4: Methotrexate, iv. Cycle 6: Venetoclax for 2 weeks,oral; Pegaspargase, im. Complete at least 6 intrathecal injections within 6 cycles.
  Interventions: Drug: Dexamethasone; Drug: Blinatumomab; Drug: Venetoclax; Drug: Inotuzumab ozogamicin; Drug: Methotrexate; Drug: Pegaspargase; Drug: Cytarabine

INTERVENTIONS:
Drug: Dexamethasone — Glucocorticoids
Drug: Blinatumomab — Bi-specific anti CD19/CD3 antibody
  Other Names: Blina
Drug: Venetoclax — BCL-2 inhibotor
  Other Names: Ven
Drug: Inotuzumab ozogamicin — a humanized monoclonal antibody-drug conjugate targeting CD22
  Other Names: INO
Drug: Methotrexate — antifolate antineoplastic drug
  Other Names: MTX
Drug: Pegaspargase — antitumor drug
  Other Names: PEG
Drug: Cytarabine — Pyrimidine, antimetabolites
  Other Names: Ara-C

SUMMARY:
Precursor B cell acute lymphoblastic leukemia (B-ALL) is an aggressive type of leukemia, with high relapse rate and poor long term survival in adults. Traditional treatment regimens mainly include chemotherapy and hematopoietic stem cell transplantation. In the past decade, with the application of molecular targeted drugs and immunotherapy, the survival of B-ALL patients has significantly improved. In this study，we propose a treatment approach that combines Blinatumomab and Venetoclax sequenced with Inotuzumab Ozogamicin in B-ALL adults. Our study aims to answer the safety and efficacy of this treatment regimen, and further improve the survival for those participants.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II and open-label study. A total of 20 Ph-negative B-ALL participants will be enrolled. The primary endpoint is 2-year event free survival(EFS).

The induction therapy is a combination of Blinatumomab(Blina), Venetoclax(Ven) and Dexamethasone(DXM), and would be applied for two cycles. As for consolidation, the Inotuzumab Ozogamicin(INO) would be given on cycle 3 and cycle 5. The high dose of MTX would be given on Cycle 4 and the Ven plus L-asp would ben given on Cycle 6. Subsequent maintenance therapy contains of low dose of Chemotherapy, Blina and INO.

The purpose of this study is to explore the safety and efficacy of the whole-process management of multi-drug combination regimen in the treatment of newly diagnosed Ph-negative B-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Before enrollment, a diagnosis of newly diagnosed precursor B-cell acute lymphoblastic leukemia with Philadelphia chromosome-negative must be confirmed. The diagnostic criteria refer to the 2022 WHO classification.
2. Age ≥ 40 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
4. Expected survival time ≥ 3 months;
5. No organ dysfunction that would restrict the use of this protocol during the screening period;
6. Understand the study and sign the informed consent form.
7. Men, women of childbearing age (only postmenopausal women who have been menopausal for at least 12 months can be considered infertile), and their partners voluntarily take effective contraceptive measures deemed effective by the investigator during the treatment period and for at least 12 months after the last dose of the study drug.

Exclusion Criteria:

1. Patients with known central nervous system (CNS) involvement of ALL;
2. Diseases with abnormal heart, lung, liver, kidney, or other organ functions that may limit the patient's participation in this trial (including but not limited to severe infections, uncontrolled diabetes, severe heart failure or angina, active pulmonary tuberculosis, asthma, COPD, bronchiectasis, etc.);
3. Cardiac ultrasound LVEF < 45%;
4. History of other malignancies within the past 5 years, excluding localized thyroid cancer and in situ skin cancer;
5. Serum total bilirubin > 1.5 ULN (upper limit of normal); ALT or AST > 2.5 ULN; serum creatinine > 1.5 ULN;
6. Known HIV infection;
7. Conditions affecting the use of the study drug as assessed by the investigator;
8. Inability to understand or comply with the study protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival(EFS) | up to 2 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first;

SECONDARY OUTCOMES:
Complete remission with or without incomplete PB cell recovery(CR/CRi) rate | at the end of Cycle 1（each cycle is 28days）
  Blast rate lower than 5% with or without peripheral blood cell recovery
Overall survival (OS) | up to 5 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of death from any cause;
Minimal residual disease (MRD) | At the end of Cycle 1（each cycle is 28 days）
  MRD level detected by flow cytometry which value <0.1% is defined as negtive

OTHER OUTCOMES:
Minimal residual disease (MRD) | At the end of Cycle 2（each cycle is 28 days）
  MRD level detected by next generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Geyer MB, Hsu M, Devlin SM, Tallman MS, Douer D, Park JH. Overall survival among older US adults with ALL remains low despite modest improvement since 1980: SEER analysis. Blood. 2017 Mar 30;129(13):1878-1881. doi: 10.1182/blood-2016-11-749507. Epub 2017 Jan 25. No abstract available. PMID 28122741
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Lu J, Zhou H, Zhou X, Yang Y, Tong L, Miao M, Yang X, Chen S. Reduced-dose chemotherapy followed by blinatumomab in induction therapy for newly diagnosed B-cell acute lymphoblastic leukemia. Cancer Med. 2024 Mar;13(5):e7062. doi: 10.1002/cam4.7062. PMID 38491815
- [Background] Kantarjian HM, DeAngelo DJ, Stelljes M, Martinelli G, Liedtke M, Stock W, Gokbuget N, O'Brien S, Wang K, Wang T, Paccagnella ML, Sleight B, Vandendries E, Advani AS. Inotuzumab Ozogamicin versus Standard Therapy for Acute Lymphoblastic Leukemia. N Engl J Med. 2016 Aug 25;375(8):740-53. doi: 10.1056/NEJMoa1509277. Epub 2016 Jun 12. PMID 27292104
- [Background] Jabbour E, Short NJ, Senapati J, Jain N, Huang X, Daver N, DiNardo CD, Pemmaraju N, Wierda W, Garcia-Manero G, Montalban Bravo G, Sasaki K, Kadia TM, Khoury J, Wang SA, Haddad FG, Jacob J, Garris R, Ravandi F, Kantarjian HM. Mini-hyper-CVD plus inotuzumab ozogamicin, with or without blinatumomab, in the subgroup of older patients with newly diagnosed Philadelphia chromosome-negative B-cell acute lymphocytic leukaemia: long-term results of an open-label phase 2 trial. Lancet Haematol. 2023 Jun;10(6):e433-e444. doi: 10.1016/S2352-3026(23)00073-X. Epub 2023 May 12. PMID 37187201